CLINICAL TRIAL: NCT04523493
Title: A Prospective, Randomized, Placebo-controlled, Double-blind, Multicenter Phase III Study to Compare Toripalimab Combined With Lenvatinib Versus Placebo Combined With Lenvatinib as the 1st-line Therapy for Advanced HCC
Brief Title: Phase III Study of Toripalimab（JS001） Combined With Lenvatinib for Advanced HCC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-027-III-HCC
Record Dates: First submitted 2020-07-09; First posted 2020-08-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Toripalimab combined with Lenvatinib
  Interventions: Combination Product: Toripalimab combined with Lenvatinib
- Control group (Placebo Comparator): Placebo combined with Lenvatinib
  Interventions: Combination Product: Placebo combined with Lenvatinib

INTERVENTIONS:
Combination Product: Toripalimab combined with Lenvatinib — Experimental group:
  Toripalimab, 240mg, IV infusion, every 3 weeks (q3w). combined with Lenvatinib 12 mg/day (Body Weight≥60 kg) or 8 mg/day (Body Weight<60 kg) oral administration, once daily. Continuous infusion, in a cycle of 3 weeks (21 days), until occurrence of termination event specified in the protocol.
  Arms: Experimental group
Combination Product: Placebo combined with Lenvatinib — Control group:
  Placebo, one unit, IV infusion, once every 3 weeks, combined with Lenvatinib 12 mg/day (Body Weight≥60 kg) or 8 mg/day (Body Weight<60 kg) oral administration, once daily. Continuous infusion, in a cycle of 3 weeks (21 days), until occurrence of termination event specified in the protocol.
  Arms: Control group

SUMMARY:
This is a prospective, randomized, placebo-controlled, double-blind, multicenter phase III registration clinical study to observe, compare and evaluate the efficacy and safety of Toripalimab combined with Lenvatinib versus placebo combined with Lenvatinib as the 1st-line therapy for advanced HCC.

Eligible subjects will be randomized at a ratio of 2:1 to receive Toripalimab combined with Lenvatinib (experimental group) or Placebo combined with Lenvatinib (control group).

ELIGIBILITY:
Inclusion criteria:

1. Age of 18-75 full years (inclusive), male or female.
2. Histopathologically or cytologically confirmed HCC or participants with liver cirrhosis meet the clinical diagnostic criteria for HCC of the American Association for the Study of Liver Diseases (AASLD).
3. Stage B (intermediate stage) or C (advanced stage) HCC determined in accordance with Barcelona Clinic Liver Cancer staging system (BCLC stage), be unsuitable for surgery and/or local therapy, or have progression of disease after surgery and/or local therapy.
4. No previous use of any systemic therapy for HCC (mainly including systemic chemotherapy, antiangiogenic drugs or other molecular targeted therapy, immunotherapy containing CTLA-4, PD 1/PD-L1 monoclonal antibody).
5. Having ≥ 1 measurable lesion in accordance with RECIST v1.1. Requirement: the selected target lesion has not been treated locally before, or is located in the area of previous local therapy and subsequently determined as PD through radiological examination and in accordance with RECIST v1.1.
6. Child-Pugh class A or ≤7 class B, with no history of hepatic encephalopathy.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score 0-1.
8. Expected survival ≥12 weeks.
9. Main organ function meets the following requirements: no blood transfusion within 14 days prior to screening, no use of hematopoietic stimulating factor (including G-CSF, GM-CSF, EPO and TPO etc.) or human albumin preparation.
10. In case of HBsAg (+) and/or HBcAb (+), HBV DNA is required to be < 1000 IU/mL (if the lowest detectable value at the local center is higher than 1000IU/mL, enrollment can be determined based on the specific condition after discussed with sponsor), and it is required to continue original anti-HBV therapy in the full course, or start to use Entecavir or tenofovir in the full course after screening during the study.
11. Female patients at childbearing age must receive serum pregnancy test within 7 days before randomization, have negative result, and are willing to use reliable and effective contraceptive methods during the trial and within 5 months after last administration. Male patients whose partners are women of childbearing potential must agree to use reliable and effective contraceptive methods during the trial and within 5 months after last administration.
12. Being voluntary to participate in the study, sufficiently informed consent and sign the written informed consent form, with good compliance.

Exclusion criteria:

1. Known cholangiocellular carcinoma (ICC) or mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma and hepatic fibrolamellar carcinoma.
2. Malignant tumor except HCC within 5 years: however, localized tumor cured in the study is excluded,including cervical carcinoma in situ, skin basal cell carcinoma and carcinoma in situ of prostate.
3. Hepatic surgery and/or local therapy or treatment with investigational product for HCC within 4 weeks prior to randomization; palliative radiation therapy for bone metastatic lesion within 2 weeks prior to randomization; use of Chinese medicine preparations with anti-liver cancer effect within two weeks prior to randomization. Toxicity induced by previous therapy (except alopecia) not recovered to ≤ grade 1 (NCI-CTCAE v5.0).
4. Prior use of other anti-PD-1 antibody or other immunotherapy targeting PD-1/PD-L1.
5. Uncontrolled pericardial effusion, uncontrolled pleural effusion or clinically obvious moderate or severe peritoneal effusion at screening, defined as reaching the following criteria: having clinical symptoms and pleural and peritoneal effusion detected in physical examination at screening; or puncture for drainage required for pleural and peritoneal effusion and/or intracavitary administration during screening.
6. History of gastrointestinal hemorrhage within 6 months prior to randomization or clear tendency of gastrointestinal hemorrhage (including severe esophageal-gastric varices with hemorrhagic risk, locally active peptic ulcer, persistent fecal occult blood (+)).
7. Having ≥ grade 3 (NCI-CTCAE v5.0) gastrointestinal or non-gastrointestinal fistula at present.
8. Cancer thrombus invasion in the main trunk of portal vein (Vp4) (more than 1/2 of the lumen), inferior vena cava cancer thrombus or cardiac involvement in accordance with CT/MRI.
9. Serious cardiovascular and cerebrovascular diseases:
10. Other obvious hemorrhagic tendency or evidence on important coagulation disorder:
11. Medium to large surgical treatment within 4 weeks prior to randomization, not including diagnostic biopsy.
12. Know central nervous system metastasis; cranial and/or spinal MRI is needed for exclusion if central nervous system metastasis is suspected.
13. Serious, uncured wound, active ulcer or untreated bone fracture.
14. Vaccination of live vaccine within 30 days prior to randomization.
15. Presence of immunodeficiency or receiving long-term systemic steroid therapy within 7 days prior to randomization (daily dose >10mg Prednisone or other equivalent glucocorticoid), or other immunosuppressive therapy.
16. Active autoimmune diseases requiring systemic treatment (i.e., immunomodulatory drug, corticosteroid or immunosuppressant) in the past two years; however, replacement therapy (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency) will not be considered as systemic therapy and is allowed to be used.
17. History of clear interstitial lung disease or non-infectious pneumonia, unless induced by local radiotherapy.
18. Active tuberculosis or received antituberculosis therapy within 1 year prior to randomization.
19. Any serious acute and chronic infection requiring systemic antibacterial, antifungal or antiviral therapy at screening, not including viral hepatitis.
20. Known history of human immunodeficiency virus (HIV) infection.
21. Previously receiving allogeneic stem cell or solid organ transplantation.
22. Inability to swallow tablets, malabsorption syndrome or any other condition that affects gastrointestinal absorption.
23. Known history of serious allergy to any monoclonal antibody, anti-angiogenesis drug.
24. Other participants who are unsuitable for inclusion as judged by the investigator."

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 3 years
  The time from randomization to death for any reason.

SECONDARY OUTCOMES:
ORR | Up to 3 years
  Defined as the proportion of subjects with the best overall response of complete response (CR) or partial response (PR).
Duration of Response (DOR) | Up to 3 years
  Defined as the time from the first evaluation of CR or PR to the first evaluation of PD or death for any reason.
DCR | Up to 3 years
  Defined as the proportion of subjects with the best overall response (BOR) of CR, PR or SD.
TTP | Up to 3 years
  Defined as the time from randomization to objective tumor progression.
Progression-free survival (PFS) | Up to 3 years
  The time from randomization to progression of disease or death for any reason, whichever comes first. Progression of disease will be evaluated
PFS rate | Up to 3 years
  The PFS rate on 6 months and 1year in both groups.
OS rate | Up to 3 years
  The OS rate on 1year and 2years in both groups.
Incidence,severity and prognosis of AEs/SAEs as assessed by NCI-CTCAE v5.0 | From date of consent informed until 90 days after the last investigational product administration. Up to 2 approximately years.
  Verbatim descriptions of adverse events will correspond to MedDRA synonymous terms, and AEs will be graded in accordance with NCI-CTCAE version 5.0. All the adverse events during or after the first dose of study drug will be summarized by treatment groups and NCI CTCAE grade. In addition, serious adverse events, adverse events (grade 3 or above) and the adverse events leading to discontinuation or suspension of study drug will be summarized correspondingly. Multiple occurrence of the same event will be counted once in accordance with the highest severity. The proportion of subjects with at least one adverse event will be reported by term of toxicity and treatment groups.
PK | To be collected once within 60 minutes prior to administration each for Toripalimab/placebo on Day 1 of Cycle (each cycle is 21 days). but the no-china sites not collection the sample
  According to the test of blood samples, the pharmacokinetic parameters of Toripalimab, mainly trough concentration, will be analyzed.
Immunogenicity | Up to 3 years
  Plasma level of anti-Toripalimab injection (JS001) antibody, immunoglobulin and Toripalimab injection (JS001) will be summarized descriptively.

OTHER OUTCOMES:
Assessment of the correlation between tumor cell PD-L1 expression level/ percentage and efficacy | Up to 3 years
  Tumor biopsy specimen collected before the treatment and tumor specimen collected at progression of tumor will be used for immunohistochemical staining test to determine the expression of PD-L1
Tumor mutation burden (TMB) | Up to 3 years
  Correlation between TMB of tumor tissue and the efficacy

CONTACTS AND LOCATIONS:
Locations (22):
- Qinhuai Medical Area, General Hospital of PLA Eastern Theater Command, Nanjing, Jiangsu, China
- Italy (5):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico,Oncologia Medica, Milan
  - IRCCS Fondazione Giovanni Pascale, Istituto Nazionale Dei Tumori, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - A.O.U. Citta della Salute e della Scienza di Torino, Tortona
  - AOUI Verona - Policlinico "G.B. Rossi" di Borgo Roma, Verona
- Poland (7):
  - Copernicus Podmiot Leczniczy sp. z o.o., Wojewodzkie Centrum Onkologii, Oddzial Onkologii Klinicznej/Chemioterapii, Gdansk
  - Szpital Wojewódzki im. Mikołaja Kopernika w Koszalinie, Oddzial Dzienny Chemioterapii, Koszalin
  - PRATIA MCM Kraków, ul. Pana Tadeusza 2,, Krakow
  - ID Clinic, Mysłowice
  - Wielkopolskie Centrum Onkologii, Oddział Onkologii Klinicznej i Immunoonkologii z Pododdziałem Dziennym i Izbą Przyjęć, Poznan
  - Centrum Medyczne Pratia Poznań, Skórzewo
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Klinika Onkologii i Radioterapii, Warsaw
- National Cancer Centre Singapore, Singapore, Singapore
- Ukraine (8):
  - Communal Non-commercial Enterprise City Clinical Hospital #4 of Dnipro City Council, Department of Chemotherapy, Dnipro
  - Communal Non-profit Enterprise "Regional Center of Oncology", Department of Abdominal Organs Oncosurgery, Kharkiv
  - Communal Non-Profit Institution of Kharkiv Regional Council Regional Clinical Specialized Dispensary of Radiation Protection of Population, Kharkiv
  - State Inst. O.O.Shalimov Nat. scientific certer of Surgery and Transplantology of Nat. Academy of Med.Sciences of Ukraine, Dep.of Oncology, Kyiv
  - Communal Enterprise Volyn Regional Clinical Hospital of Volyn Regional Council, Lutsk
  - Communal Non-commercial Enterprise Odesa Regional Clinical Hospital of Odesa Regional Council, Department of General Surgery, Odesa
  - Communal Non-commercial Enterprise of Sumy Regional Council, Sumy Regional Clinical Oncological Dispensar, Sumy
  - Communal Non-commercial Enterprise Zaporizhzhia Regional Antitumor Center of Zaporizhzhia Regional Council, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No